CLINICAL TRIAL: NCT03620669
Title: First Line Durvalumab in Patients With PD-L1 Positive, Advanced NSCLC With Performance Status 2 Unsuitable for Combination Chemotherapy. A Multicenter, Single-arm Phase II Trial
Brief Title: 1st Line Durvalumab in PS 2 NSCLC Patients
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Swiss Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SAKK 19/17
Record Dates: First submitted 2018-07-03; First posted 2018-08-08 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-08

CONDITIONS: NSCLC Stage IV; NSCLC Stage IIIB
Keywords: Lung cancer; Durvalumab; PD-L1; NSCLC; Phase II; PS 2
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms | interventions — durvalumab

STUDY DESIGN:
Intervention Model Description: Prospective single-arm open-label multicenter phase II trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Durvalumab (Experimental): Durvalumab until progression or unacceptable toxicity
  Interventions: Drug: Durvalumab

INTERVENTIONS:
Drug: Durvalumab — Durvalumab 1500mg q4W until progression or unacceptable toxicity
  Other Names: MEDI4736

SUMMARY:
The aim of the trial is to assess efficacy and safety of the treatment with durvalumab in PS 2 patients with treatment-naïve, locally advanced or metastatic, PD-L1 positive NSCLC who are considered unsuitable for combination platinum-containing therapy.

DETAILED DESCRIPTION:
Lung cancer is the leading cause of cancer deaths. An estimated 30 to 40% of patients diagnosed with NSCLC have a poor Performance status (PS) defined as a score of 2 or higher on the ECOG scale. PS 2 patients are often underrepresented in clinical trials despite representing a very frequent and important subgroup.

Platinum-based (preferably carboplatin) doublets should be considered as standard of care in eligible PS 2 patients. However the toxicity profile of platinum-based doublets remains a concern. Single-agent chemotherapy represents an alternative treatment option for the PS 2 patients considered unsuitable for platinum doublet chemotherapy but its efficacy is limited and the outcome poor.

Given the superiority of the anti-PD-1 antibody pembrolizumab versus standard chemotherapy as first line therapy in a PD-L1 positive NSCLC population, it now became the standard treatment. The PS of patients enrolled in these trials were PS 0 or 1, making the benefit of PD-L1 antibodies in PS 2 patients unclear. A retrospective real-life data analysis of nivolumab in metastatic NSCLC revealed similar treatment-related AE between patients with a PS of 0 or 1 with those having a PS of 2, confirming good treatment tolerability in poor PS patients.

The overall favorable toxicity profile of durvalumab and the absence of robust efficacy data of checkpoint inhibitors in first line treatment of patients with PD-L1 positive NSCLC with a PS of 2, encourage to investigate its activity in this cohort of patients when considered unsuitable for platinum doublet chemotherapy.

Finally, this trial aims to prolong overall survival by treating this cohort of frail patients with durvalumab, compared to historical controls, treated with single agent chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent according to Swiss law and ICH/GCP regulations before registration and prior to any trial specific procedures
* Histologically confirmed NSCLC, advanced or recurrent disease (stage IIIB to IV). Cytology could be accepted if histology is not possible
* PD-L1 expression of ≥ 25% of the tumor cells by local testing (Ventana SP142 excluded)
* No sensitizing EGFR mutation (L858R or exon 19 deletions), ALK fusion oncogene or rearrangements of the ROS1 gene detected in patients with a non-squamous cell NSCLC
* Patient unsuitable for platinum-containing combination chemotherapy according to investigator or due to patient preference
* WHO PS of 2. Confirmation of PS2 by a second medical doctor is mandatory.
* Age ≥ 18 years
* Baseline QoL forms and GA questionnaires have been completed
* Bone marrow function: hemoglobin ≥ 90 g/L, neutrophil count ≥ 1.5 x 109/L, platelet count ≥ 100 x 109/L
* Hepatic function: bilirubin ≤ 1.5 x ULN (except for patients with Gilbert's disease ≤ 3.0 x ULN); patients without liver metastases: AST and ALT ≤ 2.5 x ULN, patients with documented liver metastases: AST and ALT ≤ 5 x ULN
* Renal function: estimated glomerular filtration rate (eGFR)> 30 mL/min/1.73m² (according to CKD-EPI formula)
* Measurable or evaluable disease (by RECIST v1.1)
* Patients with asymptomatic untreated CNS metastases are eligible, provided they meet the following:

  * ≤ 5 CNS lesions with a maximum diameter of one lesion of 10 mm
  * Only supratentorial metastases allowed (i.e., no metastases to midbrain, pons, cerebellum, medulla, or spinal cord)
  * No evidence of progression at registration compared to the latest brain imaging
  * No ongoing requirement for corticosteroids as therapy for CNS disease
* Patients with symptomatic treated CNS metastases are eligible, provided they meet the following:

  * No ongoing requirement for corticosteroids as therapy for CNS disease; anticonvulsants at a stable dose allowed
  * No stereotactic radiation or whole-brain radiation within 7 days prior to registration
  * No evidence of progression at registration, after completion of CNS-directed therapy
* Tumor tissue available for central PD-L1 assessment and translational research (preferably histology but cytology could be allowed if histology is not possible). In case of scarce tumor material, a rebiopsy, if clinically possible, is encouraged
* Women with child-bearing potential are using effective contraception, are not pregnant or lactating and agree not to become pregnant during trial treatment and during the 3 months thereafter. A negative pregnancy test before inclusion into the trial is required for all women with child-bearing potential
* Men agree not to father a child during trial treatment and during 3 months thereafter
* Body weight > 30kg.
* Life expectancy > 3 months.

Exclusion criteria:

Any potential patient who meets any of the following criteria has to be excluded from entering the trial.

* History of hematologic or primary solid tumor malignancy, unless in remission for at least 3 years before registration with the exception of pT1-2 prostate cancer Gleason score <6, adequately treated cervical carcinoma in situ or localized non-melanoma skin cancer
* Prior adjuvant systemic anti-cancer treatment within 6 months before registration
* Prior systemic treatment for metastatic NSCLC
* Prior treatment with a PD-1 or PD-L1 inhibitor
* Current or prior use of immunosuppressive medication within 28 days before the first dose of durvalumab, with the exceptions of intranasal and inhaled corticosteroids or systemic corticosteroids at physiological doses (i.e. which must not exceed 10 mg/day of prednisone or an equivalent corticosteroid)
* Concomitant drugs contraindicated for use with durvalumab such as corticosteroids, methotrexate, azathioprine and tumor necrosis factor (TNF)-α blockers
* Concurrent treatment with other experimental drugs or other anticancer therapy, treatment in a clinical trial within 28 days prior to registration
* Major surgical procedure within 14 days prior to registration
* Active or prior documented autoimmune or inflammatory disorders (including inflammatory bowel disease [e.g., colitis or Crohn's disease], diverticulitis [with the exception of diverticulosis], systemic lupus erythematosus, sarcoidosis syndrome, or Wegener syndrome [granulomatosis with polyangiitis, Graves' disease, rheumatoid arthritis, hypophysitis, uveitis, etc]). The following are exceptions to this criterion:

  * Patients with vitiligo or alopecia
  * Patients with hypothyroidism (e.g., following Hashimoto syndrome) stable on hormone replacement
  * Any chronic skin condition that does not require systemic therapy
  * Patients without active disease in the last 5 years may be included but only after consultation with the coordinating investigator
  * Patients with celiac disease controlled by diet alone
* Uncontrolled diabetes mellitus
* Known history of human immunodeficiency virus (HIV) or active chronic Hepatitis C or Hepatitis B Virus infection or any uncontrolled active systemic infection requiring intravenous (iv) antimicrobial treatment
* Known history of tuberculosis
* Known history of primary immunodeficiency
* Known history of allogeneic organ transplant
* Receipt of live attenuated vaccine within 28 days prior to registration
* Severe or uncontrolled cardiovascular disease (congestive heart failure NYHA III or IV; unstable angina pectoris, history of myocardial infarction within the last six months, serious arrhythmias requiring medication (with exception of atrial fibrillation or paroxysmal supraventricular tachycardia), significant QT-prolongation, uncontrolled hypertension
* Any other serious underlying medical, psychiatric, psychological, familial or geographical condition, which in the judgment of the investigator may interfere with the planned staging, treatment and follow-up, affect patient compliance or place the patient at high risk from treatment-related complications.
* Patients with dyspnea grade ≥ 3 according to the modified Medical Research Council (mMRC) dyspnea scale.
* Patients with symptomatic pneumonitis (grade ≥ 2) or active lung infection. Patients having fully recovered from active lung infection can be included assumed they have completed antibiotics and/or corticosteroids
* Patients with disseminated intravascular coagulopathy
* Patient with a baseline CT scan older than 21 days prior to registration.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2018-12-04 (Actual); Primary Completion 2023-01-19 (Actual); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Overall survival (OS) at 6 months | At 6 months after registration
  OS at 6 months is defined as being alive at 6 months after registration.

SECONDARY OUTCOMES:
Objective response (OR) according to RECIST 1.1 | At trial treatment discontinuation or the latest 5 years after last patient discontinued trial treatment
  OR is defined as any complete response (CR) or partial response (PR) according to RECIST 1.1 criteria achieved during trial treatment.
Objective response according to iRECIST (iOR) | At trial treatment discontinuation or the latest 5 years after last patient discontinued trial treatment
  iOR is defined as any complete response (CR/iCR) or partial response (PR/iPR) according to RECIST1.1 or iRECIST criteria achieved during trial treatment.
Duration of response (DoR) according to RECIST 1.1 | At disease progression according to RECIST 1.1 criteria or death due to disease progression or the latest 5 years after last patient discontinued trial treatment
  DoR is defined as the time from the first documentation of OR until disease progression according to RECIST 1.1 criteria or death due to disease progression, whichever occurs first.
Duration of response according to iRECIST (iDoR) | At disease progression according to iRECIST criteria (iPD) or death due to disease progression or the latest 5 years after last patient discontinued trial treatment
  iDoR is defined as the time from the first documentation of iOR until disease progression according to iRECIST criteria (iPD) or death due to disease progression.
Progression-free survival (PFS) according to RECIST 1.1 | At disease progression according to RECIST v1.1 criteria or death due to any cause or the latest 5 years after last patient discontinued trial treatment
  PFS is defined as the time from registration until disease progression according to RECIST v1.1 criteria or death due to any cause, whichever occurs first.
Progression-free survival according to iRECIST (iPFS) | At disease progression according to iRECIST criteria (iPD) or death due to any reason or the latest 5 years after last patient discontinued trial treatment
  iPFS is defined as the time from registration until disease progression according to iRECIST criteria (iPD) or death due to any reason, whichever occurs first.
  iPD is defined as the time point of first iUPD without subsequent iSD, iPR or iCR before trial treatment discontinuation.
  Patients not experiencing an event at the time of the analysis, as well as patients starting a subsequent anticancer treatment in the absence of an event, will be censored at the date of their last available tumor assessment showing no evidence of iPD before starting a subsequent anticancer treatment, if any.
Overall survival (OS) | At death of the patient or the latest 5 years after last patient discontinued trial treatment
  OS is defined as the time from registration until death due to any cause
Adverse events (AEs) | From registration until 28 days after last trial treatment dose
  All AEs will be assessed according to NCI CTCAE v5.0
Quality of life (QoL): Core 30 (QLQ-C30) | From registration until trial treatment discontinuation or the latest 1 year after registration
  QoL is measured by the Questionnaire Core 30 (QLQ-C30) including the complementary Lung Cancer Module (QLQ-LC13)
Geriatric assessment (GA) - Screening instrument (G8) | At baseline
  Screening instrument (G8)
Geriatric assessment (GA) - Assessment with IADL | At baseline
  Assessment with IADL
Geriatric assessment (GA) | At baseline
  Comorbidities assessment with CCI

CONTACTS AND LOCATIONS:
Overall Officials: Michael Mark, MD, Study Chair — Kantonsspital Graubünden
Locations (11):
- Switzerland (11):
  - Kantonsspital Aarau, Aarau
  - Kantonsspital Baden, Baden
  - Universitaetsspital Basel, Basel
  - IOSI Ospedale Regionale di Bellinzona e Valli, Bellinzona
  - Inselspital, Bern
  - Kantonsspital Graubuenden, Chur
  - Hopital Fribourgeois HFR, Fribourg
  - Hôpitaux Universitaires de Genève, Geneva
  - Kantonsspital - St. Gallen, Sankt Gallen
  - Spital STS AG, Thun
  - Kantonsspital Winterthur, Winterthur